CLINICAL TRIAL: NCT05817864
Title: Diagnostic Accuracy of Using Capnography in Verification of Nasogastric Tube Placement in Hospital Settings
Brief Title: Diagnostic Accuracy of Capnography in Nasogastric Tube Placement
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Chau Pak Chun Janita, Professor, Chinese University of Hong Kong
Other Study IDs: 2022073
Record Dates: First submitted 2023-03-23; First posted 2023-04-18 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Capnography; Nasogastric Tube; Diagnostic Accuracy
Keywords: Capnography; Intubation, gastrointestinal; Diagnostic accuracy
MeSH Terms: interventions — Capnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational group: All participants included will be in one observational cohort.
  Interventions: Diagnostic Test: Capnography

INTERVENTIONS:
Diagnostic Test: Capnography — Index test: Capnography, which monitors ETCO2, the percentage concentration, or partial pressure of CO2 at the end of exhalation, will serve as the index test. It will be performed by connecting the end of the nasogastric tube with the sensor of the bedside sidestream capnography device. Placement within the airway is defined as detecting a capnogram waveform or an ETCO2 level > 10 mmHg.
  Reference standard: This study will use radiography (chest/abdominal X-ray) as the reference standard for determining the correct placement of nasogastric tubes. Radiology will be performed as soon as possible and interpreted by a physician. A repeat radiography will be performed if necessary. We will also use pH-Fix-4.5-10 to determine the pH value, and its accuracy is +/- 0.2 pH with minimum increments of 0.5. A pH of 5.5 or below indicates gastric placement.

SUMMARY:
A prospective observational diagnostic study will be conducted to assess the sensitivity and specificity of using capnography in detecting the correct placement of nasogastric tubes using the reference standards of radiography and measurement of aspirates for pH value.

DETAILED DESCRIPTION:
A prospective observational diagnostic study will be conducted. Patients ≥ 18-year-old and requiring the insertion of an nasogastric tube will be recruited using a convenience sampling method from general medical and geriatric wards, intensive care units (ICUs), accident and emergency departments (AEDs), and subacute/rehabilitation/infirmary wards in 21 acute or subacute/convalescent/extended care hospitals. End-tidal carbon dioxide (ETCO2) detection by sidestream capnography, which indicates airway intubation of an nasogastric tube when a capnogram waveform or an ETCO2 level > 10 mmHg, will serve as the index test. The reference standards will be the pH value of gastric content aspiration (pH ≤ 5.5 indicates gastric placement) and X-ray performed after the index test. Each participant will be included only once. Sensitivity, specificity, positive predictive value, and negative predictive value, and the area under the receiver operating characteristic curve of capnography will be calculated to assess the diagnostic performance of capnography. The variability in diagnostic accuracy in participants with different characteristics will be compared. The time spent and the cost of the index test and the reference test will be compared.

This study will provide evidence on the diagnostic accuracy of capnography in verifying nasogastric tube placement and inform the update of clinical practice guidelines and stakeholders' decisions regarding the adoption of ETCO2 detection as a routine method for verifying nasogastric tube placement.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or above;
* Admitted to the general medical and geriatric wards, ICUs, or subacute/rehabilitation/infirmary wards in subacute/convalescent/extended care hospitals or visiting AEDs in acute hospitals;
* Requiring the insertion of an nasogastric tube into the stomach for assessment, nutritional support and medication administration during the study period.

Exclusion Criteria:

* Participants receiving life-saving intervention at the time of recruitment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A convenience sampling method will be adopted in this study. The participants will be recruited from general medical and geriatric wards, ICUs, AEDs, and subacute/rehabilitation/infirmary wards in 21 acute or subacute/convalescent/extended care hospitals. Each participant will be included in the study once.
Sampling Method: Non-Probability Sample
Enrollment: 390 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of Capnography | Through study completion, an average of 2 year
  True Positive / (True Positive + False Negative) × 100%
Specificity of Capnography | Through study completion, an average of 2 year
  True Negative / (True Negative + False Positive) × 100%
Positive Predictive Value of Capnography | Through study completion, an average of 2 year
  True Positive / (True Positive + False Positive) × 100%
Negative Predictive Value of Capnography | Through study completion, an average of 2 year
  True Negative / (True Negative + False Negative) × 100%
Overall diagnostic performance of Capnography | Through study completion, an average of 2 year
  Measured by the area under the receiver operating characteristic curve (AUROC). The test accuracy level is considered high when the AUROC value is ≥ 0.9.

SECONDARY OUTCOMES:
Difference in the time spent of index test and reference test | Through study completion, an average of 2 year
  Compare the time spent of index test (i.e., capnography) and reference test (i.e., radiography)
Difference in the cost of index test and reference test | Through study completion, an average of 2 year
  Compare the cost of index test (i.e., capnography) and reference test (i.e., radiography)

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong SAR, China

IPD SHARING:
Plan to Share IPD: No
The datasets generated during and/or analysed during the current study will be available from the principal investigator on reasonable request.

REFERENCES:
- [Background] Chau JP, Thompson DR, Fernandez R, Griffiths R, Lo HS. Methods for determining the correct nasogastric tube placement after insertion: a meta-analysis. JBI Libr Syst Rev. 2009;7(16):679-760. doi: 10.11124/01938924-200907160-00001. PMID 27820026
- [Background] Chau JP, Lo SH, Thompson DR, Fernandez R, Griffiths R. Use of end-tidal carbon dioxide detection to determine correct placement of nasogastric tube: a meta-analysis. Int J Nurs Stud. 2011 Apr;48(4):513-21. doi: 10.1016/j.ijnurstu.2010.12.004. Epub 2011 Jan 7. PMID 21215969
- [Background] Chau JPC, Liu X, Choi KC, Lo SHS, Lam SKY, Chan KM, Zhao J, Thompson DR. Diagnostic accuracy of end-tidal carbon dioxide detection in determining correct placement of nasogastric tube: An updated systematic review with meta-analysis. Int J Nurs Stud. 2021 Nov;123:104071. doi: 10.1016/j.ijnurstu.2021.104071. Epub 2021 Aug 24. PMID 34520886
- [Derived] Chau JPC, Tong DWK, Lo SHS, Sze SYM, Kwok MLM, Lai PCK, Lam HKC, Chung JYM, Liu X, Chien WT, Choi KC. Diagnostic accuracy of using capnography in verification of nasogastric tube placement among adult patients in hospital settings: Protocol of a diagnostic study. PLoS One. 2023 Oct 23;18(10):e0292667. doi: 10.1371/journal.pone.0292667. eCollection 2023. PMID 37871102